CLINICAL TRIAL: NCT02689505
Title: Phase I, Non-randomized, Open-label, Multi-center Dose Escalation Trial of BI 836880 Administered by Weekly Repeated Intravenous Infusions in Patients With Advanced Solid Tumors.
Brief Title: Weekly BI 836880 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1336.6; 2015-001132-38 (EudraCT Number)
Record Dates: First submitted 2016-02-23; First posted 2016-02-24 (Estimated); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (5):
- 40 mg BI 836880 (Experimental): 40 mg BI 836880
  Interventions: Drug: BI 836880
- 120 mg BI 836880 (Experimental): 120 mg BI 836880
  Interventions: Drug: BI 836880
- 150 mg BI 836880 (Experimental): 150 mg BI 836880
  Interventions: Drug: BI 836880
- 180 mg BI 836880 (Experimental): 180 mg BI 836880
  Interventions: Drug: BI 836880
- 240 mg BI 836880 (Experimental): 240 mg BI 836880
  Interventions: Drug: BI 836880

INTERVENTIONS:
Drug: BI 836880 — Solution for intravenous infusion

SUMMARY:
This is a Phase I, multi-centre, non-randomized, uncontrolled, open-label, dose escalating study of BI 836880 administered intravenously once a week. The eligible patient population will be patients with advanced solid tumors.

The primary objective of this trial is to determine the maximum tolerated dose (MTD) and recommended Phase II doses for BI 836880 in patients with solid tumors. Preliminary safety data will be evaluated as secondary objectives.

Subsequently, pharmacokinetic profile, pharmacodynamic changes in circulating biomarkers and Dynamic Contrast-Enhanced Magnetic Resonance Imaging ( DCE-MRI), anti-tumor activity and the immunogenicity of BI 836880 will be explored up to a total of 40 patients with advanced solid tumors.

Dose escalation will be guided by a Bayesian logistic regression model with over dose control (EWOC) using at least 2 patients per dose cohorts.

Safety criteria will be followed, including adverse events according to Common Terminology Criteria (CTCAE version 4.03), incidence of dose limiting toxicities, physical examination, vital signs, safety laboratory parameters and Eastern Cooperative Oncology Group (ECOG).

ELIGIBILITY:
Inclusion criteria:

1 Age >=18 years 2. Histologically confirmed malignancy which is locally advanced or metastatic solid tumor, and either refractory after standard therapy for the disease or for which standard therapy is not reliably effective e.g. patients do not tolerate or have contraindications to otherwise available standard therapy and tumour lesions evaluable for Dynamic contrast-enhanced (DCE)-MRI at MTD.

3. ECOG performance status <= 2 4. Adequate hepatic, renal and bone marrow functions as defined by the following criteria:

1. Total bilirubin within normal limits (<= 1.5x upper limit of normal (ULN) for patient with Gilberts syndrome)
2. Alanine amino transferase (ALT) and aspartate amino transferase (AST) <= 1.5x ULN (< 5x upper limit of normal (ULN) for patient known liver metastases)
3. Serum creatinine < 1.5x ULN
4. International normalized Ratio (INR) 0.8-1.2 or partial thromboplastin time (PTT) < 1.5x ULN
5. Absolute neutrophil count (ANC) > 1.5 109/L
6. Platelet count > 100x109/ L.
7. Haemoglobin > 10 g/dl (without transfusion within previous week) 5. Signed and dated written informed consent. 6. Life expectancy >= 3 months in the opinion of the investigator 7. Recovery from all reversible adverse events of previous anti-cancer therapies to baseline or CTCAE grade1, except for alopecia (any grade), sensory peripheral neuropathy CTCAE grade <= 2 or considered by the investigator as clinically not significant.

   8. Male or female patients. Women of childbearing potential* must be ready and able to use highly effective methods of birth control per International Conference on Harmonisation [ICH M3(R2)] in combination with male condom as "double barrier", during the trial and for at least 6 months after the end of treatment with BI 836880, that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.

   Male patient must always use condoms when sexually active during the trial and for at least 6 months after the end of treatment with BI 836880.

   *Women of childbearing potential are defined as: Any female who has experienced menarche and does not meet the criteria for "women not of childbearing potential" as described below.

   Women not of childbearing potential are defined as:

   Women who are postmenopausal (12 months with no menses without an alternative medical cause) or who are permanently sterilized (e.g., hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

   Exclusion criteria:
   1. Known hypersensitivity to the trial drugs or their excipients or risk of allergic of anaphylactic reaction to the study drug according to the investigator judgement (e.g. patient with history of anaphylactic reaction or autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs (NSAIDS), inhaled corticosteroids, or the equivalent of < 10 mg/day prednisone)
   2. Current or prior treatment with any systemic anti-cancer therapy either within 28 days or a minimum of 5 half-lives, whichever is shorter at the start of study treatment.
   3. Serious concomitant disease (based on investigator judgement), especially those affecting compliance with trial requirements or which are considered relevant for the evaluation of the endpoints of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the investigator would make the patient inappropriate for entry into the trial.
   4. Major injuries and/or surgery (as judged by the investigator) or bone fracture within 4 weeks of start of study treatment, or planned surgical procedures during the trial period.
   5. Patients with personal or family history of QT prolongation and/or long QT syndrome, or prolonged QT interval corrected for heart rate according to Fridericia's formula (QTcF) at baseline (> 470 ms). QTcF will be calculated by Investigator as the mean of the 3 ECGs taken at screening.
   6. Significant cardiovascular/ cerebrovascular disease (i.e uncontrolled hypertension, unstable angina, history of infarction within past 6 months, congestive heart failure > New York heart association ( NYHA II). Uncontrolled hypertension defined as: blood pressure in tested and relaxed condition >= 140 mmHg, systolic or > 90 mmHg diastolic (with or without medication), measured according to Section 5.3.2 and Appendix 10.2.
   7. History of severe haemorrhagic or thromboembolic event in the past 12 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis).
   8. Known inherited predisposition to bleeding or to thrombosis in the opinion of the investigator.
   9. Patient with brain metastases that are symptomatic and/or require therapy.
   10. Patients who require full-dose anticoagulation (according to local guidelines). No vitamin K antagonist and other anticoagulation allowed; low-molecular-weight heparin (LMWH) allowed only for prevention not for curative treatment.
   11. Use of alcohol or drug incompatible with patient participation in the study in the investigator opinion
   12. Patient unable or unwilling to comply with protocol
   13. Women who are pregnant, nursing, or who plan to become pregnant while in the trial
   14. Previous enrolment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- CTR Georges-François Leclerc, Dijon, France
- Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Derived] Keller S, Kunz U, Schmid U, Beusmans J, Buchert M, He M, Jayadeva G, Le Tourneau C, Luedtke D, Niessen HG, Oum'hamed Z, Pleiner S, Wang X, Graeser R. Comprehensive biomarker and modeling approach to support dose finding for BI 836880, a VEGF/Ang-2 inhibitor. J Transl Med. 2024 Oct 14;22(1):934. doi: 10.1186/s12967-024-05612-x. PMID 39402675
- [Derived] Le Tourneau C, Becker H, Claus R, Elez E, Ricci F, Fritsch R, Silber Y, Hennequin A, Tabernero J, Jayadeva G, Luedtke D, He M, Isambert N. Two phase I studies of BI 836880, a vascular endothelial growth factor/angiopoietin-2 inhibitor, administered once every 3 weeks or once weekly in patients with advanced solid tumors. ESMO Open. 2022 Oct;7(5):100576. doi: 10.1016/j.esmoop.2022.100576. Epub 2022 Sep 13. PMID 36108560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, non-randomised, uncontrolled, dose-escalating trial in patients with advanced solid tumors.
Pre-assignment Details: All subjects who were screened for eligibility to participate in the trial signed informed consent. Subject were assigned to the trial drug if the met all the inclusion and none of the exclusion criteria.
  Abbreviations: AE = Adverse Event.
Groups:
- 40 mg BI 836880: 40 milligram (mg) solution of BI 836880 was administered as once weekly intravenous infusion in 3 weeks treatment cycles. Participants continued treatment until disease progression or unacceptable toxicity.
- 120 mg BI 836880: 120 mg solution of BI 836880 was administered as once weekly intravenous infusion in 3 weeks treatment cycles. Participants continued treatment until disease progression or unacceptable toxicity.
- 150 mg BI 836880: 150 mg solution of BI 836880 was administered as once weekly intravenous infusion in 3 weeks treatment cycles. Participants continued treatment until disease progression or unacceptable toxicity.
- 180 mg BI 836880: 180 mg solution of BI 836880 was administered as once weekly intravenous infusion in 3 weeks treatment cycles. Participants continued treatment until disease progression or unacceptable toxicity.
- 240 mg BI 836880: 240 mg solution of BI 836880 was administered as once weekly intravenous infusion in 3 weeks treatment cycles. Participants continued treatment until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 150 mg BI 836880 | 180 mg BI 836880 | 240 mg BI 836880
Started | 2 | 5 | 3 | 11 | 3
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 5 | 3 | 11 | 3
Not completed — Progressive disease | 2 | 2 | 3 | 9 | 1
Not completed — Dose Limiting Toxicity | 0 | 1 | 0 | 0 | 2
Not completed — Other AE or clinical progression | 0 | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All patients who were treated with at least one single dose of BI 836880.
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 150 mg BI 836880 | 180 mg BI 836880 | 240 mg BI 836880 | Total
Number analyzed (Participants) | 2 | 5 | 3 | 11 | 3 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.0 (15.6) | 61.8 (9.7) | 56.0 (22.1) | 56.0 (12.6) | 62.0 (4.6) | 57.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 7 | 2 | 17
  Male | 1 | 1 | 0 | 4 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 7 | 2 | 14
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 4 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Determination of the maximum tolerated dose (MTD) in participants with advanced solid tumors. MTD was defined as the highest dose with less than 25% risk of true DLT rate being above 33% in the MTD evaluation period, and could be considered reached if the probability that the true DLT rate was in the target interval (16% to 33%) was sufficiently large during the MTD evaluation period. The MTD evaluation period was defined as 3 weeks after first administration of treatment.
Time Frame: First treatment cycle, 3 weeks from first administration of trial treatment (MTD evaluation period).
Population: Dose-finding cohort treated set: All patients enrolled in dose finding and confirmation of MTD cohort of the trial who were documented to have taken at least 1 dose of trial medication and were evaluable for MTD determination.
Measure: Number; unit: Milligram (mg)
Groups:
- Total BI 836880: Participants were administered 40/ 120/ 150 / 180 /240 milligram (mg) solution of BI 836880 as once weekly intravenous infusion in 3 weeks treatment cycles. Participants continued treatment until disease progression or unacceptable toxicity.
Arm/Group | Total BI 836880
Number analyzed (Participants) | 19
Milligram (mg) | 180

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in the Maximum Tolerated Dose (MTD) Evaluation Period
Description: The following drug-related adverse events qualified as DLTs: Common Terminology Criteria for Adverse Events (CTCAE) grade 4 neutropenia >7 days or complicated by infection; grade >3 febrile neutropenia; grade = 4 thrombocytopenia; grade > 3 thrombocytopenia with bleeding; grade > 3 proteinuria > 3 non haematological toxicity except: Vomiting or diarrhea responding to supporting treatment, fatigue lasting for less than 4 days, transient grade 3 infusion reaction, any laboratory abnormality, which was considered not clinically relevant by the investigator or resolved spontaneously or could be resolved with appropriate treatment. Hypertension: increase of diastolic blood pressure (BP) by 15 mmHg, which could not be controlled by hypertensive medication and requires a dose reduction of BI 836880 for further treatment course. All related AE leading to an interruption of BI 836880 for more than 14 days until recovery to baseline.
Time Frame: First treatment cycle, 3 weeks from first administration of trial treatment (MTD evaluation period).
Population: Dose finding cohort treated set: All patients enrolled in dose finding and confirmation of MTD cohort of the trial who were documented to have taken at least 1 dose of trial medication and were evaluable for the MTD determination.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 150 mg BI 836880 | 180 mg BI 836880 | 240 mg BI 836880 | Total BI 836880
Number analyzed (Participants) | 2 | 5 | 3 | 6 | 3 | 19
Participants | 0 | 1 | 0 | 1 | 2 | 4

3. Secondary Outcome: Number of Participants With Drug-related Adverse Events (AEs) Leading to Dose Reduction or Discontinuation During the Treatment Period
Description: Number of Participants with drug-related adverse Events (AEs) leading to dose reduction or discontinuation during the treatment period.
Time Frame: From first trial drug administration until 42 (Residual Effect Period) days after the last trial drug administration, up to 566 days.
Population: Treated Set: The treated set includes all participants enrolled in the Trial who were documented to have taken at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 150 mg BI 836880 | 180 mg BI 836880 | 240 mg BI 836880 | Total BI 836880
Number analyzed (Participants) | 2 | 5 | 3 | 11 | 3 | 24
Participants | 0 | 3 | 0 | 1 | 2 | 6

ADVERSE EVENTS:
Time Frame: From first trial drug administration until 42 (Residual Effect Period) days after the last trial drug administration, up to 566 days.
Description: Treated set: All participants who were treated with at least one single dose of BI 836880.
Arm/Group | 40 mg BI 836880 | 120 mg BI 836880 | 150 mg BI 836880 | 180 mg BI 836880 | 240 mg BI 836880 | Total BI 836880
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5 | 0/3 | 0/11 | 0/3 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/2 | 3/5 | 0/3 | 6/11 | 2/3 | 12/24
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5 | 3/3 | 11/11 | 3/3 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg BI 836880 (N=2) | 120 mg BI 836880 (N=5) | 150 mg BI 836880 (N=3) | 180 mg BI 836880 (N=11) | 240 mg BI 836880 (N=3) | Total BI 836880 (N=24)
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg BI 836880 (N=2) | 120 mg BI 836880 (N=5) | 150 mg BI 836880 (N=3) | 180 mg BI 836880 (N=11) | 240 mg BI 836880 (N=3) | Total BI 836880 (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1 | 6
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 4
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1 | 5
Asthenia (General disorders) | 2 | 4 | 1 | 7 | 1 | 15
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 1 | 0 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 2 | 0 | 3
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Xerosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 2
Stoma site erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 3 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 3 | 0 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
QRS axis abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 2 | 2 | 0 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 0 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 4
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 1 | 4
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1
Vulval oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 0 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 3
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review Prior to any Submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI´s intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT02689505/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT02689505/SAP_001.pdf